CLINICAL TRIAL: NCT01483560
Title: Phase 3 Study of Metformin in Adults With Type 1 Diabetes
Brief Title: REducing With MetfOrmin Vascular Adverse Lesions in Type 1 Diabetes (REMOVAL)
Acronym: REMOVAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); Juvenile Diabetes Research Foundation (Other); Imperial College London (Other); University of Wisconsin, Madison (Other); University of Dundee (Other); Merck Serono S.A., Geneva (Industry); Itamar-Medical, Israel (Industry); University of Western Ontario, Canada (Other); University of Melbourne (Other); Steno Diabetes Center Copenhagen (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Prof John Petrie, Clinical Professor in Diabetic Medicine, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GN10DI406; 2011-000300-18 (EudraCT Number)
Record Dates: First submitted 2011-11-23; First posted 2011-12-01 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: REMOVAL; metformin; carotid IMT; LDL Cholesterol; endothelial function; retinopathy; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Retinal Diseases | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Oral Metformin (as Glucophage 500mg x 2 bd) titrated from initial 500mg to target 2000mg daily
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 3 years treatment duration
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — 3 years duration
  Arms: Placebo

SUMMARY:
The trial is conducted in the United Kingdom (UK), Australia, Canada, Denmark and the Netherlands. The aim is to test whether 3 years treatment with metformin added to titrated insulin therapy (towards target HbA1c 7.0%/53 mmol/mol) reduces atherosclerosis, as measured by progression of carotid intima-media thickness (cIMT), in adults with confirmed type 1 diabetes aged 40 years and over at increased risk for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes for five years or more*
* Age 40 years or above
* 7.0 =< HbA1c <10.0% (53 - 86 mmol/mol)

AND 3 or more of the following ten CardioVascular Disease (CVD) risk factors:

* BMI >27 kg/m^2
* Current HbA1c >8.0% (64 mmol/mol)
* Known CVD/peripheral vascular disease
* Current smoker
* Estimated glomerular filtration rate (eGFR) <90 ml/min per 1.73 m^3
* Confirmed micro- or macroalbuminuria [according to local assays and reference ranges]
* Hypertension (BP >=140/90 millimeters of mercury (mmHg) or established on antihypertensive treatment)
* Dyslipidaemia [total cholesterol >=5.0 mmol/L (200 mg/dL);OR HDL cholesterol <1.20 mmol/L (46mg/dL) [MEN]; OR <1.30 mmol/L (50 mg/dL) [WOMEN]; or triglycerides >=1.7 mmol/L (150mg/dL); or established on lipid-lowering treatment)]
* Strong family history of CVD (at least one parent, biological aunt/ uncle, or sibling with myocardial infarction or stroke aged <60 years)
* Duration of diabetes > 20 years

Exclusion Criteria:

* eGFR < 45 ml/min/1.73m2
* woman of childbearing age not on effective contraception
* Pregnancy and/or lactation
* Acute coronary syndrome or Stroke/Transient Ischaemic Attack within the last three months
* NYHA stage 3 or 4 heart failure
* Significant hypoglycaemia unawareness
* Impaired cognitive function/ unable to give informed consent
* Previous carotid surgery/ inability to capture adequate carotid images
* Estimated glomerular filtration < 45ml/min/1.73m^2 (MDRD)
* Gastroparesis
* History of lactic acidosis
* Other contraindications to metformin (hepatic impairment, known hypersensitivity to metformin, acute illness such as dehydration, severe infection, shock, acute cardiac failure or suspected tissue hypoxia)
* Any coexistent life threatening condition including prior diagnosis of cancer within two years
* History of alcohol problem or drug abuse

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2011-12; Primary Completion 2017-03-19 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Petrie, Prof, Principal Investigator — University of Glasgow; Helen Colhoun, Prof, Study Director — University of Dundee
Locations (24):
- Australia (3):
  - Royal Melbourne Hospital, Melbourne
  - St Vincent's Hospital, Melbourne
  - Royal Prince Albert Hospital, Sydney
- Canada (2):
  - St Joseph's Health Care, London, Ontario
  - Ottawa Hospital Riverside Campus, Ottawa
- Steno Diabetes Centre, Gentofte Municipality, Denmark
- Maastricht University Medical Centre, Maastricht, Netherlands
- United Kingdom (17):
  - Aberdeen Royal Infirmary, Aberdeen
  - Ayr Hospital, Ayr
  - University Hospitals Bristol, Bristol
  - Diabetes Support Unit, Ninewells Hospital and Medical School, Dundee
  - University Hospital North Durham, Durham
  - Edinburgh Royal Infirmary, Edinburgh
  - Edinburgh Western Infirmary, Edinburgh
  - Peninsula NIHR Clinical Research Facility, Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Stobhill Hospital, Diabetes Clinic, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Michael White Diabetes Centre, Hull Royal Infirmary, Hull
  - Clinical Sciences Centre, University Hospital, Liverpool
  - Clinical Investigation Unit, International Centre for Circulatory Health, Imperial College Healthcare NHS Trust, London
  - Wellcome Trust Clinical Research Facility, Manchester Royal Infirmary, Manchester
  - Newcastle NIHR Clinical Research Facility, Royal Victoria Hospital, Newcastle
  - Diabetes Clinical Research Centre, Plymouth, Plymouth
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: Yes
Site specific participant data will be made available to the site PIs later in 2017, after the main publications.

REFERENCES:
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240
- [Derived] Petrie JR, Chaturvedi N, Ford I, Brouwers MCGJ, Greenlaw N, Tillin T, Hramiak I, Hughes AD, Jenkins AJ, Klein BEK, Klein R, Ooi TC, Rossing P, Stehouwer CDA, Sattar N, Colhoun HM; REMOVAL Study Group. Cardiovascular and metabolic effects of metformin in patients with type 1 diabetes (REMOVAL): a double-blind, randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2017 Aug;5(8):597-609. doi: 10.1016/S2213-8587(17)30194-8. Epub 2017 Jun 11. PMID 28615149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 493 participants where enrolled and consented. All participants entered a 3 month Run In phase with placebo. Participants who remained eligible were randomly assigned to receive metformin or placebo for 3 years. 65 participants where ineligible to be randomized.
Groups:
- Metformin: Oral Metformin (as Glucophage 500mg x 2 bd) titrated from initial 500mg to target 2000mg daily
  Metformin: 3 years treatment duration 219 of 428 randomised were assigned to Metformin Group
- Placebo: Placebo: 3 years duration 209 of the 428 randomised were assigned to Placebo
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 219 | 209
Completed | 193 | 194
Not Completed | 26 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 219 | 209 | 428
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 219 | 209 | 428
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (8.5) | 55.8 (8.8) | 55.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 85 | 175
  Male | 129 | 124 | 253
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 55 | 55 | 110
  Netherlands | 16 | 15 | 31
  Denmark | 4 | 4 | 8
  United Kingdom | 112 | 105 | 217
  Australia | 32 | 30 | 62
Diabetes Diagnosis Duration [Mean (Standard Deviation); unit: years] | 33.4 (11) | 34.3 (10.5) | 33.85 (10.75)
Existing Cardiovascular Disease [Number; unit: participants] | 30 | 22 | 52
Baseline HbA1c [Number; unit: mmol/mol] | 64.8 | 64.7 | 64.75
Daily Insulin Dose [Number; unit: units/kg] | 0.63 | 0.68 | 0.66
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.4 (4.5) | 28.5 (4.1) | 28.5 (4.3)
Blood Pressure [Mean (Standard Deviation); unit: Systolic BP (mmHg)] | 130.5 (15) | 128.5 (14.6) | 129.5 (14.8)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4 (0.88) | 4 (0.93) | 4 (0.91)
eGFR [Mean (Standard Deviation); unit: ml/min/1.73m2] | 92.9 (20.9) | 91.1 (21.6) | 92 (21.3)
Diabetic Retinopathy [Number; unit: participants] | 51 | 58 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change in Averaged Mean Far Wall Common Carotid Artery Intima-media Thickness (cIMT)
Description: Progression of averaged mean far wall common carotid artery intima media thickness IMT (mean cIMT) measured using B mode ultrasonography with a 7.0 MHz or higher broadband linear array transducer and concurrent recording of 3-lead electrocardiogram (ECG). Longitudinal images of the common carotid artery will be obtained at anterior, lateral and posterior angles at baseline, 12, 24 and 36 months using Meijer's arc to standardize the transducer angle.
Time Frame: 0, 12 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 193 | 194
mm
  Baseline | 0.773 (0.14) | 0.791 (0.183)
  12 Months | 0.782 (0.147) | 0.788 (0.174)
  24 Months | 0.792 (0.145) | 0.823 (0.187)
  36 Months | 0.793 (0.134) | 0.820 (0.177)

2. Secondary Outcome: Change in HbA1c
Description: Measured in accredited local laboratories participating in DCCT-aligned quality control programmes.
Time Frame: Baseline, Year 3
Measure: Mean (Standard Deviation); unit: %units
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 193 | 194
%units
  Baseline | 8.1 (0.9) | 8.0 (0.8)
  36 Months | 8.1 (0.9) | 8.1 (0.8)

3. Secondary Outcome: Change in LDL Cholesterol
Description: mmol/L Centrally assayed at the University of Glasgow
Time Frame: Baseline, Year 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 193 | 194
mmol/L
  Baseline | 2.23 (0.7) | 2.25 (0.72)
  36 Months | 2.07 (0.83) | 2.21 (0.71)

4. Secondary Outcome: Change in Estimated Glomerular Filtration Rate
Description: Number of participants developing new microalbuminuria; change in absolute concentration Calculated using the MDRD equation1 based on creatinine measured in accredited local laboratories
Time Frame: Baseline, Year 1, Year 2, Year 3
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 193 | 194
ml/min/1.73m2
  Baseline | 92.9 (20.9) | 91.1 (21.6)
  36 Months | 92.1 (20.8) | 87.2 (19.6)

5. Secondary Outcome: Number of Participants With Retinopathy and at Least a 2 Stage Progression in Retinopathy From Baseline to 36 Months
Description: Two color 45° field retinal photographs (fields 1 and 2) from each eye at 0 and 36 months graded at the University of Wisconsin Ocular Epidemiology Reading Center (OERC) using the modified Airlie House classification scheme and the Early Treatment Diabetic Retinopathy Severity scale.
Time Frame: Baseline, Year 3
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 219 | 209
Participants
  Baseline | 191 | 190
  36 Months | 8 | 10

6. Secondary Outcome: Change in Weight
Description: Measured at sites using calibrated weighing scales
Time Frame: Baseline, Year 1, Year 2, Year 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 193 | 194
kg
  Baseline | 83.9 (15.4) | 83.5 (13.7)
  36 Months | 82.0 (15.4) | 83.2 (13.8)

7. Secondary Outcome: Change in Insulin Dose
Description: Units/ kg body weight Extracted by study nurses from the Study Diary and reported on the study CRF using dedicated fields
Time Frame: Baseline, Year 1, Year 2, Year 3
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 193 | 194
units/kg
  Baseline | 0.36 (0.26) | 0.68 (0.30)
  36 Months | 0.62 (0.26) | 0.67 (0.30)

8. Secondary Outcome: Change in Endothelial Function
Description: In some centres (Arbitrary units) Reactive Hyperaemia Index using the ENDOPAT device (Itamar, Israel)
Time Frame: Baseline, Year 1, Year 3
Measure: Mean (Standard Deviation); unit: RHI (Arbitrary units)
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 193 | 194
RHI (Arbitrary units)
  Baseline | 2.28 (0.74) | 2.24 (0.75)
  36 Months | 2.17 (0.69) | 2.24 (0.73)

ADVERSE EVENTS:
Time Frame: Adverse event data collected from the date of consent until 30 days post last IMP dose, an average of 3 years.
Description: Definition used same as clinical trials.gov
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 5/219 | 2/209
Serious Adverse Events (participants affected / at risk) | 34/219 | 31/209
Other Adverse Events (participants affected / at risk) | 112/219 | 52/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=219) | Placebo (N=209)
Metabolic and nutrition (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Infections and Infestations (Infections and infestations) | 7 (7) | 5 (5)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 4 (4) | 5 (5)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Cardiac (Cardiac disorders) | 3 (3) | 6 (6)
Injury (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Coronary artery bypass graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Angiogram (Investigations) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Blood and Lymphatic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune System Disorder (Immune system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
hypoglycaemic coma (Nervous system disorders) | 1 (1) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
lung lobectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
coronary stent insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Amputation revision (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgery (unspecified) (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal fusion Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic valve repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Blood Glucose Fluctuation (Investigations) | 0 (0) | 1 (1)
Ischaemic Necrosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=219) | Placebo (N=209)
Gastrointestinal (Gastrointestinal disorders) | 88 (88) | 18 (18)
Cardiovascular (Cardiac disorders) | 1 (1) | 1 (1)
Neurological (Nervous system disorders) | 0 (0) | 0 (0)
Hypersensitivity to Metformin (Product Issues) | 5 (5) | 1 (5)
Opthalmic adverse events (Eye disorders) | 18 (18) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT01483560/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT01483560/SAP_001.pdf